CLINICAL TRIAL: NCT02589743
Title: Impact of the Intermediary Layer on Sealant Retention: A Randomized 24-month Clinical Trial
Brief Title: Randomized Clinical Trial of Occlusal Sealant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Profa. Dra. Regina Maria Puppin Rontani, Teacher, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1
Record Dates: First submitted 2015-10-17; First posted 2015-10-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Dental Caries
Keywords: clinical trial; pit and fissure sealants; tooth eruption; retention; adhesive system; intermediary layer
MeSH Terms: conditions — Dental Caries; Van der Woude syndrome; Exanthema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fluroshield - F (Sealant) (Active Comparator): Pit and fissure sealing using only sealant
  Interventions: Device: Sealant
- Single Bond and F (Adhesive and Sealant) (Experimental): Pit and fissure sealing using adhesive and sealant
  Interventions: Device: Adhesive and Sealant
- Helioseal Clear Chroma - H (Sealant) (Active Comparator): Pit and fissure sealing using only sealant
  Interventions: Device: Sealant
- Excite and H (Adhesive and Sealant) (Experimental): Pit and fissure sealing using adhesive and sealant
  Interventions: Device: Adhesive and Sealant

INTERVENTIONS:
Device: Sealant — Application of preventive agent
  Arms: Fluroshield - F (Sealant); Helioseal Clear Chroma - H (Sealant)
Device: Adhesive and Sealant — Application of preventive agent and technique for control moisture
  Arms: Excite and H (Adhesive and Sealant); Single Bond and F (Adhesive and Sealant)

SUMMARY:
This study assessed long-term impact of tooth Eruption Stages (ES) on sealant retention on occlusal surfaces previously coated with intermediary bonding layer and it determined caries incidence outcome evolved. The treatment were (sealant/technique): Fluroshield; Helioseal Clear Chroma; Single Bond and Fluroshield; Excite and Helioseal Clear Chroma.

DETAILED DESCRIPTION:
The greatest risk of sealant failure occurs soon after tooth eruption, when contamination with saliva and gingival fluid is almost inevitable. The use of an intermediate bonding layer between humidity contaminated enamel and sealant can improve bond strength, reduces microleakage, and enhances resin flow into fissures. The benefit of primer and adhesive layer beneath the sealant seems to be based on a combination of moisture-chasing effects of the hydrophilic primer, increased flow dispersion imparted by the less viscous primer and adhesive and increased flexibility of the combined and polymerized primer/adhesive/resin complex once reaction is complete.

ELIGIBILITY:
Inclusion Criteria:

* Four caries-free erupted first molar permanent teeth; no systemic diseases and no dental material allergies.

Exclusion Criteria:

* Carious or absence first molar permanent teeth.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2003-04; Primary Completion 2003-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Sealant retention and prevention of dental caries assessed by defined clinical scoring system | 6-mouth
  Clinical scoring system: adapted criteria proposed by Feigal et al. (2000)

CONTACTS AND LOCATIONS:
Overall Officials: Kamila Kantovitz, Phd, Principal Investigator — Piracicaba Dental Scholl - University of Campinas; Kelly Moreira, DDS, Principal Investigator — Piracicaba Dental Scholl - University of Campinas